CLINICAL TRIAL: NCT06950788
Title: Changes in Glucose Tolerance in Patients With Cirrhosis Peri-Liver Transplant
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-0691
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cirrhosis, Liver; Diabetes Mellitus Risk; Transplant; Failure, Liver; Transplant-Related Disorder
Keywords: Cirrhosis; Post-transplant diabetes; New-onset diabetes after transplant; Liver transplantation
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected will include blood, urine, and stool. If the subject goes to liver transplant, during the surgery tissue will be collected from the implanting liver, explant liver, abdominal muscle, visceral fat, and subcutaneous fat. If the subject obtains a standard of care liver biopsy, an extra pass may be taken for liver tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to establish risk factors for post-transplant in adult individuals with cirrhosis without diabetes undergoing liver transplant evaluation.

The question being addressed is: can laboratory work, anthropometric tests, functional tests, imaging, and advanced measurements such as wrist actigraphy, continuous glucose monitoring, or oral glucose tolerance testing predict the development of diabetes after liver transplant?

Participants will be asked to periodically participate in wearing a continuous glucose monitor and wrist actigraph and obtain an oral glucose tolerance test both before and after liver transplant.

DETAILED DESCRIPTION:
Participants will be enrolled from the liver transplant clinic and will be given a continuous glucose monitor, a wrist actigraph, a home sleep apnea testing device, and a questionnaire packet to collect demographics, sleep quality, and physical activity information. They will be scheduled for an outpatient two-hour oral glucose tolerance test, which will use a frequently sampling protocol to allow for mathematical modeling of insulin secretion. They will undergo body composition measurements using a bio-electrical impedance analysis device. Subjects will undergo these tests, excluding the home sleep apnea test, every three months until and through liver transplantation, after which they will restart the protocol at three months, or one month after post-transplant steroids are weaned to their lowest level. After they are one year post-transplant, they will no longer participate in continuous glucose monitoring or oral glucose tolerance testing, but their care will be followed electronically to assess outcomes up to five years post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to liver transplant clinic with a diagnosis of cirrhosis.
* Age >18 yrs.
* Ability to understand and sign written consent form, or have a legally-authorized representative or proxy who can be approached for consent

Exclusion Criteria:

* Patients without consent
* Patients with implantable cardioverter defibrillator devices or automated implantable cardioverter defibrillator devices will be excluded from the bio-electrical impedance analysis portion of the measurements.
* Patients with unremovable electrical medical devices or devices that cannot turn off will be excluded from the bio-electrical impedance analysis measurements
* Pregnant patients
* Incarcerated patients
* Patients with a history of type 2 diabetes mellitus diagnosed > 5 years ago will be excluded from the Oral Glucose Tolerance Test portion of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with cirrhosis undergoing evaluation for liver transplant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Early post-transplant hyperglycemia | 45 days after transplant
  Blood sugars above 200 mg/dL or requiring insulin therapy
Post-transplant diabetes | 45 days to 365 days after liver transplant
  Hemoglobin A1c > 6.5% or two-hour glucose from an oral glucose tolerance test ≥ 200 mg/dL after liver transplant

SECONDARY OUTCOMES:
Undiagnosed diabetes in cirrhosis | Before transplant
  Two-hour glucose in an oral glucose tolerance test ≥ 200 mg/dL in an individual with cirrhosis with a hemoglobin A1c less than 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Rinella, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No